CLINICAL TRIAL: NCT02412683
Title: Neurotoxic Symptoms in Adjuvant Chemotherapy in Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Jenny Drott (Other Government)
Responsible Party: Sponsor-Investigator, Jenny Drott, RN, Ph-D student, Linkoeping University
Organization: Linkoeping University (Other Government)
Other Study IDs: NTOX-123
Record Dates: First submitted 2015-01-16; First posted 2015-04-09 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: oxaliplatin

SUMMARY:
Subgroups of patients with radically operated colorectal cancer can have a better prognosis by over six months are treated with chemotherapy. This beneficial effect may be enhanced somewhat by providing a combination of chemotherapy and the addition of oxaliplatin. It is known that this treatment additions increase the risk of neurotoxic side effects such as sensitivity to cold, numbness and tingling in hands or feet, muscle cramps, pain, taste disorders and swallowing difficulties.

The aim is to investigate how colorectal cancer patients with oxaliplatin adjuvant chemotherapy experience neurotoxic effects and if the experience of the symptoms change over time during treatment and how symptoms affect patients' daily lives and quality of life.

DETAILED DESCRIPTION:
Subgroups of patients with radically operated colorectal cancer can have a better prognosis by over six months are treated with chemotherapy. This beneficial effect may be enhanced somewhat by providing a combination of chemotherapy and the addition of oxaliplatin. It is known that this treatment additions increase the risk of neurotoxic side effects such as sensitivity to cold, numbness and tingling in hands or feet, muscle cramps, pain, taste disorders and swallowing difficulties. A few studies on patients' experience of the neurotoxic symptoms and its impact on daily life.

The operative treatment of colorectal cancer is surgery. The possibility of curative resection is the factor most strongly associated to the patient's survival. High-risk patients and metastasis is not a contraindication for surgery of the primary tumor, but the individual patient's benefit from surgery must be especially valued. If the primary tumor does not cause any troublesome symptoms, and there are metastases in other organs, which can be treated with non-surgical methods, the tumor can be left initially and removed later if symptoms occur. For rectal cancer radiation therapy can be topical and reduces the risk of local recurrence. In locally advanced cancer in which radical resection is not possible, radiation therapy, with or without chemotherapy, be current in order to achieve tumor-killing effect of the infiltration zone. Radiation therapy can cause acute and chronic complications, such as pain, faecal incontinence and sexual dysfunction which may affect patients' quality of life.

At more advanced but radically operated colorectal cancer is commonly advised chemotherapy. The goal of giving chemotherapy is that, if possible, prevent micrometastasis that may exist in any patient, even though the patient is managed with radical surgery. Colorectal cancer spreads primarily to the lymph nodes and liver, but also through the bloodstream to the lungs, brain and bone. Choice of chemotherapy is influenced by several factors, including tumor extent, time from primary diagnosis, previous treatment given, symptoms, performance status, concomitant other diseases, blood tests and patient's own attitude towards such readiness to accept some side effects. Treatment intention can be curative, palliative or prophylactic (adjuvant). There are mainly three types of chemotherapy used to treat colorectal cancers. They can be individual, but is usually provided in combination. They can be given in multiple lines, which means that a combination can be administered initially and then changed to another combination of poor tolerance or treatment failure. Most patients get two or three lines of treatment.

Intended to provide combination therapy is to increase efficacy against the tumor, reducing the risk of resistance developing and spreading side effects. The effect of a particular treatment is best the earlier it is given but may be meaningful even at a later stage. A cornerstone of treatment for over five decades, 5-fluorouracil (5FU), which in colorectal cancer, in combination with folinic acid (leucovorin). This regime is relatively lowtoxic and most patients are capable of treatment without severe side effects. Capecitabine (Xeloda) is another treatment regimen, which is often preferred by patients because it is given orally and usually mild side effects. Another treatment option is to give oxaliplatin in addition to 5-flurouracil, leucovorin or capecitabine (FOLFOX 4, PHLOX, XELOX). These combinations are under trials to prolong survival compared with only 5-flurouracil and leucovorin. Oxaliplatin can reduce the risk of relapse by about 25 percent in comparison with 5FU/leukovorin. This regimen poses an increased proportion of neurotoxic side effects as a result. Chemotherapy can generally provide a number of unpleasant and sometimes life-threatening side effects. Side effects that may occur are symptoms of nausea, vomiting, diarrhea, anemia, skin lesions and mouth blown.

This can result in nutritional difficulties, reduced strength and impaired immune system with increased risk of infection.

The fact that the patient be informed of a cancer diagnosis is a strain on both the patient but also for the relatives. This may mean that ordinary life is changing and that the normal daily activities can not be performed previously because of hospitalization, surgical and oncological treatment. As far as quality of life as it includes the experience of health and welfare of the patient based on physical, psychological and social needs. It may also include economic, political, and spiritual needs. The concept of health-related quality of life suited to the context in which disease symptoms affect the individual's physical function. Possible treatments and its side effects can affect individual's ability to function. Health-related quality of life is an individual experience and can vary between individuals. In the case of the most valuable views on the treatment results so the patient has a very important role. Patients who have a disease with a reading experience both advantages and disadvantages (side effects) with their treatment. By measuring the patients' health-related quality of life it is possible to create a picture of the patient's perspective on their illness and treatment.

Sense Of Coherence (SOC) has been by Antonovsky divided into three key components: comprehensibility, manageability and meaningfulness. Antonovsky argues that the degree of SOC affects a person's ability to handle stressful situations. Studies show that psychological stress has a negative impact on quality of life in patients with various types of cancer, but few studies have shown that the same applies to colorectal cancer patients. But the cancer patients' personality affects the perceived quality of life is known. Several psychological and personality factors play a central role in the disease process. A strong sense of coherence is a health-stimulating factor and in studies of cancer patients resulted in reduced mortality, disease progression and resignation. The cancer involves the patient an extensive psychological stressful situation, and the patient's capacity to adapt themselves to be influenced by his defense. The validated instrument SOC (Sense of Coherence) is able to measure the patients' sense of coherence.

Neurotoxic side effects often occur during treatment with oxaliplatin. Oxaliplatin can cause acute and delayed neuropathies. Studies have shown that some patients have persistent and chronic problems. Acute neurotoxicity is usually a half hour to an hour after start of infusion and disappears after a few days, and often arrives at any doses. These symptoms can present themselves as paresthesia, cold intolerance, and pain in the eye and jaw, abdominal pain, cramps in legs and calves, numbness and tingling of the hands, feet and around his mouth and voice and vision changes. Side effects are not reduced within 14 days can be permanent nerve damage leading to difficulties to write, walk, swallow and carry out daily activities. Permanent damage may occur without acute side effects initial stage. It is important that especially during the second half of the treatment period, observe signs of neurotoxic symptoms consisting of therapy. Studies show that the neurotoxic effects greatly affected how long the treatment lasted. If patients have these side effects should oxaliplatin reduced or excluded for fear debilitating and prolonged neuropathy.

The drug-specific questionnaire Oxaliplatin-Specific Neurotoxicity Scale is the most accurate instrument for measuring the neurotoxic symptoms. The instrument is divided into three parts: upper extremities, lower extremities and mouth / facial region. Symptoms estimated from the preceding cycle of therapy and graded based on whether symptoms exist or not. If the patient has symptoms, these should be graded from 1-5. Patients should also rate the extent to which symptoms affect their daily lives and activities between 1-5.

It is important to note early neurotoxic effects and to encourage patients to report symptoms that arise. Information before treatment is started if the side effects that might arise and how patients can detect early symptoms are significant.

Patients who had neuropathy in the upper extremities experienced difficulties such as fastening buttons, zips close, write, sew and do housework, unlike the patients with lower neuropathy who had difficulty driving, walking, train and carry out activities (balance). The perceived disability can cause feelings of anxiety, depression, frustration, anger and difficulty in adapting to their situation which may also affect the social interaction.

The aim is to investigate how colorectal cancer patients with oxaliplatin adjuvant chemotherapy experience neurotoxic effects and if the experience of the symptoms change over time during treatment and how symptoms affect patients' daily lives and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients recieved adjuvant oxaliplatin chemotherapy after radical surgery
* Ability to answer questions in swedish language
* Ability to answer questions in mobile telephone

Exclusion Criteria:

* Colorectal cancer patients in other regimes (palliative setting, no surgery)
* Non ability to answer questions in swedish language
* Non ability to answer questions in mobile telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients recieved adjuvant oxaliplatin chemotherapy after radical surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Oxaliplatin-Specific Neurotoxicity Scale | up to 12 months

SECONDARY OUTCOMES:
Health related quality of life (Fact-G) Questionnaire | up to 12 months
Sense of Coherence scale (SOC-scale) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carina Bertero, RN,professor, Study Director — Department of Health Sciences
Locations (1):
- Jenny Drott, Linköping, Sweden

REFERENCES:
- [Derived] Drott J, Fomichov V, Borjeson S, Bertero C. Sense of coherence and health-related quality of life in patients with neurotoxicity after cancer chemotherapy: Assessment from a real-time mobile phone-based system. Psychooncology. 2020 Jan;29(1):107-113. doi: 10.1002/pon.5243. Epub 2019 Oct 31. PMID 31670431